CLINICAL TRIAL: NCT06106581
Title: A Randomized, Observer-blinded, Dose Response Phase 2 Trial to Assess the Safety and Immunogenicity of Two Different Dose Levels of a Live-attenuated Chikungunya Virus Vaccine (VLA1553) in Healthy Children Aged 1 to 11 Years
Brief Title: A Phase 2 Clinical Trial of VLA1553 in Healthy Children Aged 1 to 11 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA1553-221
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- VLA1553 full dose (Experimental)
  Interventions: Biological: VLA1553 full dose
- VLA1553 half dose (Experimental)
  Interventions: Biological: VLA1553 half dose
- Control (Active Comparator): Single intramuscular vaccination on Day 1 with Nimenrix (Men ACWY vaccine), a conjugate vaccine indicated for the active immunization
  Interventions: Biological: Control

INTERVENTIONS:
Biological: VLA1553 full dose — Single intramuscular vaccination on Day 1 with VLA1553 full dose, a lyophilized live-attenuated Chikungunya vaccine candidate
  Arms: VLA1553 full dose
Biological: VLA1553 half dose — Single intramuscular vaccination on Day 1 with VLA1553 half dose, a lyophilized live-attenuated Chikungunya vaccine candidate
  Arms: VLA1553 half dose
Biological: Control — Nimenrix
  Arms: Control

SUMMARY:
This is a multicenter, prospective, randomized, observer-blinded, three arm, phase 2 clinical trial evaluating the full dose formulation of VLA1553, half dose formulation of VLA1553 and control.

At least 300 male and female healthy children aged 1 to 11 years will be enrolled and the overall distribution of participants will be 2:2:1 to the two VLA1553 dose groups (n=120 each) or control (n=60).

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, observer-blinded, three arm, phase 2 clinical trial evaluating the full dose formulation of VLA1553, half dose formulation of VLA1553 and control (Nimenrix, a tetravalent meningococcal vaccine - Men ACWY).

At least 300 male and female healthy children aged 1 to 11 years will be enrolled and the overall distribution of participants will be 2:2:1 to the two VLA1553 dose groups (n=120 each) or control (Nimenrix) (n=60).

As a safety precaution measure, the first 30 sentinel participants will be enrolled into the trial in an open-label fashion according to an age step down scheme.

After sentinel analysis, participants will be enrolled in a blinded, randomized manner into three Trial Arms. Within each treatment arm participants will be stratified into three age strata:

Stratum A: 7 to 11 years -children from their 7th birthday until the day before their 12th birthday.

Stratum B: 3 to 6 years - children from their 3rd birthday until the day before their 7th birthday.

Stratum C: 1 to 2 years - children from their 1st birthday until the day before their 3rd birthday.

Age strata for the VLA1553 treatment arms are targeted to be equal in size, i.e., approximately 40 per age stratum.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy children aged 7 to 11 years for Stratum A, 3 to 6 years for Stratum B and 1 to 2 years for Stratum C at the time of vaccination;
2. Written informed consent by the participant's parent(s)/Legally Acceptable Representative(s) ((LAR(s)), according to local requirements, and written informed assent of the participant, if applicable;

Exclusion Criteria:

1. Participant who is IgM+/IgG- does not qualify for participation in this trial.
2. Participant is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical trial involving an investigational CHIKV vaccine;
3. Participant has an acute or recent infection (and who is not symptom-free in the week prior to the Screening Visit (Visit 0)

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited injection site reactions | within 14 days post-vaccination
Severity of solicited injection site reactions | within 14 days post-vaccination
Frequency of systemic reactions | within 14 days post-vaccination
Severity of systemic reactions | within 14 days post-vaccination

SECONDARY OUTCOMES:
Frequency of any adverse event (AE) | within 28 days post-vaccination
Severity of any adverse event (AE) | within 28 days post-vaccination
Frequency of unsolicited AE | until Month 6 (Day 180) and Month 12 (Day 365) post-vaccination
Severity of unsolicited AE | until Month 6 (Day 180) and Month 12 (Day 365) post-vaccination
Frequency of any serious adverse event (SAE) | until Month 6 (Day 180) and Month 12 (Day 365) post-vaccination
Severity of any serious adverse event (SAE) | until Month 6 (Day 180) and Month 12 (Day 365) post-vaccination
Immune response in baseline seronegative participants as measured by CHIKV-specific neutralizing antibody titers | on Day 1, Day 15, Day 29, Day 85, Day 180 and Month 12 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (3):
- Dominican Republic (2):
  - Fundacion Dominicana de Perinatologia Fundacion Probebe, Santo Domingo, Gazcue
  - Instituto Dermatologico y Cirugia de la Piel "Dr Huberto Bogaert Diaz" IDCP, Santo Domingo
- Inversiones en Investigacion Medica INVERIME, Tegucigalpa, Honduras

IPD SHARING:
Plan to Share IPD: Yes
After trial completion, Valneva may provide access to individual de-identified participant data and related trial documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Trial Report (CTR)) upon request from qualified researchers, and subject to Valneva's review and approval.

REFERENCES:
- [Derived] Weisova P, Scheiblauer S, Ecker J, Schneider M, Hochreiter R, Bitzer A, Kosulin K, Schoengrundner P, Fuchs U, Rodeles L, Mazara S, Donastorg Y, Rivera S, Wressnigg N, Dubischar K, Buerger V, Eder-Lingelbach S, Jaramillo JC. Live-attenuated chikungunya vaccine in children: a randomized phase 2 trial. Nat Med. 2026 Feb 6. doi: 10.1038/s41591-025-04197-2. Online ahead of print. PMID 41652122